CLINICAL TRIAL: NCT02322008
Title: Anti-TNF Therapy in Danish Patients With Inflammatory Bowel Diseases in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Regionshospitalet Viborg, Skive (Other)
Responsible Party: Principal Investigator, Steffen Bank, M.sc, phd, Regionshospitalet Viborg, Skive
Other Study IDs: Anti-TNF, IBD
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Infliximab; Adalimumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: infliximab and adalimumab — In this retrospective, observational study, no interventions were undertaken by the researchers.
  Other Names: remicade and humira, anti-TNF

SUMMARY:
Can genetic markers be used to predict anti-TNF response? A cohort was established to identify SNPs associated with anti-TNF therapy in patients with inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* CD or UC, treated with anti-TNF

Exclusion Criteria:

* Missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1035 patients with CD or UC
Sampling Method: Non-Probability Sample
Enrollment: 1035 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
3-step scale | 22 weeks
  Best response within 22 weeks

REFERENCES:
- [Derived] Bank S, Andersen PS, Burisch J, Pedersen N, Roug S, Galsgaard J, Turino SY, Brodersen JB, Rashid S, Avlund S, Olesen TB, Green A, Hoffmann HJ, Thomsen MK, Thomsen VO, Nexo BA, Vogel U, Andersen V. Effectiveness of anti-tumour necrosis factor-alpha therapy in Danish patients with inflammatory bowel diseases. Dan Med J. 2015 Mar;62(3):A4994. PMID 25748864